CLINICAL TRIAL: NCT02901119
Title: Effects of Whey Protein Consumption by Patients Waiting for Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CAAE-27430714.8.0000.5149
Record Dates: First submitted 2016-02-04; First posted 2016-09-15 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2016-09

CONDITIONS: Liver Disease; Nutrition Disorders
MeSH Terms: conditions — Liver Diseases; Nutrition Disorders | interventions — Whey Proteins; Caseins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whey protein (Experimental): Patients are instructed to consume 20g of whey protein in the morning and 20g at night, during 15 days, as a supplement. Their regular usual diet is maintained.
  Interventions: Dietary Supplement: Whey protein
- Casein (Active Comparator): Patients are instructed to consume 20g of casein in the morning and 20g at night, during 15 days, as a supplement. Their regular usual diet is maintained.
  Interventions: Dietary Supplement: Whey protein

INTERVENTIONS:
Dietary Supplement: Whey protein — Patients, maintaining their regular usual diet, are submitted to a protein supplementation, during 15 days. They recieve 20g packages of whey protein or casein, to take twice a day: 20g in the morning and 20g at night.
  Other Names: Casein

SUMMARY:
Malnutrition is prevalent among chronic liver disease patients. Inadequate ingestion and/or metabolic alterations modify the body composition and biological functions. The purpose of this study is to determine whether whey protein comsumption, due to amino acid profile, digestibility and bioactive compounds may be beneficial for patients waiting for liver transplantation

DETAILED DESCRIPTION:
A randomized, double-blind, intervention study in which patients are randomly assigned to receive packages of 20g of whey protein (WP) or casein (CA) to take twice a day (20g in the morning and 20g at night), as a supplement, during 15 days. They are monitored weekly by calls. Regular usual diet is maintained. Patients underwent muscle functionality assessment by handgrip dynamometry and 6-min. walking test and, the inflammatory response by plasmatic cytokines. All tests are performed at the beginning and the end of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Chronic liver disease, liver transplantation

Exclusion Criteria:

* Children, illiterate, elderly, renal failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | Two years
  Anthropometry
Nutritional status | Two years
  Functionality - dynometry

SECONDARY OUTCOMES:
Heart rate variability | Two years
  Heart rate variability
Resting energy expenditure | Two years
  Calorimetry

CONTACTS AND LOCATIONS:
Locations (1):
- UFMG Hospital, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No